CLINICAL TRIAL: NCT01365104
Title: Hypoxia-Inducible Transcription Factor 1 (HIF-1)in Vascular Aging
Brief Title: Modulation of Cerebral Blood Flow Using Iron Chelators
Acronym: DFO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Farzaneh Sorond, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1K23AG030967-01 (NIH); 1K23AG030967-01A1 (NIH)
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Stroke; Problem of Aging
Keywords: brain blood flow; stroke; cerebrovascular; aging; cerebrovascular hemodynamics
MeSH Terms: conditions — Stroke | interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy young (Experimental): Each subject comes for 2 visits. There is a randomized, double-blind, crossover design so each subject will receive active drug during one visit and placebo during the other.
  Interventions: Drug: desferrioxamine
- healthy old (Experimental): Each subject comes for 2 visits. There is a randomized, double-blind, crossover design so each subject will receive active drug during one visit and placebo during the other.
  Interventions: Drug: desferrioxamine

INTERVENTIONS:
Drug: desferrioxamine — intravenous infusion at 10mg/kg/hr for a total of 6 hours at final infused doses of 60mg/kg.
  Other Names: Desferal, desferoxamine

SUMMARY:
The purpose of this study is determine if the iron chelator, desferrioxamine can increase blood levels of hypoxia-inducible transcription factor 1 (HIF-1 protein) and to see if there is a corresponding increase in blood flow to the brain.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults between the ages of 18-80 years.

Exclusion Criteria:

* subjects taking vasoactive medications,
* hypertension,
* pregnant women, smokers,
* COPD,
* asthma,
* diabetes mellitus,
* intracranial or carotid stenosis,
* hepatic disease,
* renal disease,
* bone marrow suppression,
* cardiac disease,
* heart failure,
* iron deficiency,
* history of cancer,
* history of head trauma,
* subarachnoid hemorrhage,
* central nervous system vasculitis,
* multiple sclerosis,
* migraines,
* seizures,
* sickle cell disease or trait,
* cardiac arrhythmia,
* unable to give informed consent, or
* poor transcranial Doppler insonation windows.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Define change from baseline cerebral blood flow after receiving DFO infusion. | baseline, 3hr, 6hr, 9hr
  Cerebral blood flow is measured with transcranial Doppler ultrasound at baseline and then study drug is initiated. Blood flow is measured again after 3 hours of infusion, 6 hours of infusion, then once more 3 hours after the infusion is complete.
Determine if DFO changes blood HIF-1 levels from baseline and whether this correlates with changes in cerebrovascular hemodynamics. | baseline, 3hr, 6hr, 9hr
  Blood samples are taken at each time point and will be correlated with ultrasound blood flow measures taken at baseline, 3hrs of infusion, 6hrs of infusion, and 3 hours after infusion is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh Sorond, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sorond FA, Tan CO, LaRose S, Monk AD, Fichorova R, Ryan S, Lipsitz LA. Deferoxamine, Cerebrovascular Hemodynamics, and Vascular Aging: Potential Role for Hypoxia-Inducible Transcription Factor-1-Regulated Pathways. Stroke. 2015 Sep;46(9):2576-83. doi: 10.1161/STROKEAHA.115.009906. Epub 2015 Jul 30. PMID 26304864